CLINICAL TRIAL: NCT01641003
Title: Isolation and Characterization of Cancer Stem Cells Using iFP Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: cancer stem cells.ctil
Record Dates: First submitted 2012-06-26; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Neoplasm of Breast; Glioma; Pancreatic Cancer
Keywords: cancer stem cells
MeSH Terms: conditions — Breast Neoplasms; Glioma; Pancreatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of fresh tumors taken after surgery without compromising final histology diagnosis. These specimens will be used to isolate and grow cancer stem cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fresh tumor specimen: Fresh tumor specimen taken immediately after surgery of patients diagnosed with pancreatic cancer, GBM and Breast cancer. These specimens will be taken immediately to the lab isolate and grow CSC using the described methods. No specific intervention done regarding the patients- the samples taken will be processed in the lab.

SUMMARY:
1. to evaluate insoluble fibrinogen particles (iFP), as a tool for harvesting, growing and transferring attachment-dependent cancer stem cells and comparing it to the standard method ( coated plate) .
2. to evaluate whether using iFP for growing CSC can yield better results of isolating and enriching CSCs from fresh tumors than other conventional methods

DETAILED DESCRIPTION:
There has been a growing interest in recent years on cancer stem cells (CSC) and their implication in cancer biology and therapy.

CSCs refer to a subset of tumor cells that has the ability to self-renew and generate the diverse cells that comprise the tumor.

These cells have been termed cancer Stem cells to reflect their 'stem-like' properties and ability to continually initiate and sustain tumorigenesis.

CSCs share important properties with normal tissue stem cells, including self-renewal (by symmetric and asymmetric division) and differentiation capacity, albeit aberrant. Multilineage differentiation, however, is not a mandatory feature of a CSC. Furthermore, these cells are thought to be resistant to conventional cancer therapy including chemotherapy and radiotherapy which may explain rapid tumor cell repopulation following treatment mainly by this subtype of cells, therefore new therapeutic method to target CSCs are now under thorough investigation.

One of the major difficulties in finding and identifying CSC is that they are hard to isolate, grow, and enrich.

Several in vitro assays have been used to identify stem cells, including sphere assays, serial colony-forming unit (CFU) assays (replating assays), and label-retention assays.

Studies have also been performed with the goal of determining genetic signatures that define CSCs. However, each of these methods has potential pitfalls that complicate interpretation of the results.

Therefore additional method to easily harvest and enrich the CSCs is required. Currently, the vast majority of cells are cultivated in 2-D flat hard plastic plates and flasks that are inert to the cells. However CSCs are grown in a 3-D serum free conditions which make their growth slow and complicated.

Often proteins, such as fibronectin or collagen, have been employed as coatings to render the plastic more "cell friendly". However yields are still low; costs are high, and require much floor space (large footprint). Moreover, the cells attached to the plastic must be trypsinized in order to transfer or to implant affecting the survival of cells exposed to digesting enzymes.

Fibrinogen is an acute phase protein , occurring at 2-4g/l in human blood, upon treatment with glucocorticoid, inflammation or trauma, the concentration of fibrinogen increase Fibrinogen exerts adhesive effect on cultured fibroblast and other cells. Specifically fibrinogen and its various lytic fragments (D.E ,FPA )were shown to be chemotactic to macrophage , human fibroblast and endothelial cells.

Fibrin matrix is commonly used surgical hemostasis and tissue sealing Fibrin(ogen) - a possible candidate from which a 3-D matrix for cell culturing could be fabricated, is the major component of the blood coagulation system. Native fibrinogen is soluble in aqueous buffer and cannot usually be employed for cell culture applications, except as a coating for plastics. However, when mixed with a trace of thrombin, it becomes transformed into an insoluble fibrin clot that attracts cells and provides a provisional matrix for tissue repair.

Experimental plan:

1. Generating and enriching CSC (in vitro) from established cell lines of human cancer We will isolate, purify, and characterize CSC from a series of established cell line including , U87-MG human glioma, MCF7 breast carcinoma and PANC-1 human pancreatic adenocarcinoma, using standard techniques as described in Methods . These cells will be cultured and grown as monolayer's in serum containing medium or as spheres in serum free medium supplemented by growth factors .(18-7-19) We will evaluate the ability of the cells to form spheres and characterize their stem cell properties using surface markers detection and measuring ALDH activity.
2. Growing CSCs on iFP substance:

   iFP may exhibit high attachment response for cancer cells, conserve cell surface marker, and yield optimal growth rate. In addition, the cells on IFP could be transferred without trypsinization which can diminish cell damage during harvesting from plastic plate resulting in higher survival.

   Cells will be cultured in dishes coated iFP substance as described in the Methods. After 2 weeks in culture, cells will be harvested identified for CSCs for cancer stem cell proprieties using the same methods we described above (e.g surface markers and ALDH activity) .
3. To isolate and enrich CSCs from fresh tumor specimens This aim designed to promote the implication of iFP in cancer research by studying, harvesting, and growing CSCs obtained from fresh tumors and subsequently using them for in vitro therapeutic testing. Such an approach can optimize the therapy which may target this type of cell.

Tumor specimens will be obtained from consenting patients according to the Internal Review and The Ethics Board.

Tumor samples will be collected from the pathology department from the histological diagnostic assessment during tumor resection (when the samples are still fresh). Thus samples will be received in the Laboratory within 30 minutes of surgery.

Tumors will be prepared as single cell suspensions and then will be grown using either conventional standard method or iFP. Subsequently, cells will be harvested and evaluated for CSC characteristics using the same method we used for cell lines. A comparison of the yield of CSC percentage will be performed between iFP and the conventional methodology.

ELIGIBILITY:
Inclusion Criteria:

1. Above 18 years old.
2. Signed ICF.
3. Expected to under go cancer removing surgery in Rambam MC.
4. A sample of the tumor can be brought to the lab within 30 of its removal.
5. Enough histological material to perform a good histological evaluation.

Exclusion Criteria:

1. Patient not interested to participate in clinical trial.
2. PI decision.
3. Chemotherapy or radiotherapy treatment prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with GBM, Pancreas or Breast cancer who are planed to undergo surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Cancer stem cells percentage | 24 months
  Evaluation of CSCs and non-CSCs population by using several surface markers. For glioma and pancreas, CSC are defined as CD133 positive. For breast carcinoma CSCs are identified as CD44+/CD24-/Low. Percentage of CSCs will be measured for comparing the yield of the methods using iFP and the standard method.

CONTACTS AND LOCATIONS:
Overall Officials: FADI - MIZYED, Dr., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel